CLINICAL TRIAL: NCT00661635
Title: A Multiple-Dose, Randomized, Double-Blind, Placebo-Controlled Study of the Analgesic Efficacy and Safety of Valdecoxib Compared to Placebo in Patients for Treatment of Post-Surgical Pain From Laparoscopic Cholecystectomy Surgery
Brief Title: A Randomized, Double-Blind Study of the Efficacy and Safety of Valdecoxib Compared to Placebo for Treatment of Post- Cholecystectomy Surgery Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VALA-0513-145; A3471085
Record Dates: First submitted 2008-03-31; First posted 2008-04-18 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-03

CONDITIONS: Laparoscopic Cholecystectomy; Pain
Keywords: Laparoscopic Cholecystectomy Surgery, Acute Pain, Perioperative Pain
MeSH Terms: conditions — Pain; Acute Pain | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — valdecoxib 40 mg by mouth within 8 hours after the end of surgery, followed by a second dose of valdecoxib 20 mg within 1 to 12 hours (or by midnight on the Day 1, whichever was earlier); then, placebo twice daily (BID) on Days 2 to 5
  Arms: Arm 3
Drug: valdecoxib — valdecoxib 40 mg by mouth within 8 hours after the end of surgery, followed by a second dose of valdecoxib 20 mg within 1 to 12 hours (or by midnight on the Day 1, whichever was earlier); then, valdecoxib 20 mg once daily (QD)on Days 2 to 5.
  Arms: Arm 2
Drug: valdecoxib — valdecoxib 40 mg by mouth within 8 hours after the end of surgery, followed by a second dose of valdecoxib 20 mg within 1 to 12 hours (or by midnight on the Day 1, whichever was earlier); then, valdecoxib 20 mg twice daily (BID) on Days 2 to 5.
  Arms: Arm 1

SUMMARY:
To evaluate the analgesic efficacy, general safety, and effects on health outcome measures and opioid-related symptoms of 2 valdecoxib dosing regimens compared with placebo in patients with moderate or severe pain following laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients had required an elective, non-urgent laparoscopic cholecystectomy, as an outpatient procedure, with ASA Class I-III, with a Baseline Pain Intensity of moderate or severe on a categorical scale and ≥45 mm on a VAS (100 mm)
* Patients were able to get their first dose of study medication within 8 hours after the end of surgery

Exclusion Criteria:

* Patients could not undergo procedures expected to produce a greater degree of surgical trauma than the laparoscopic cholecystectomy alone, nor have acute pre-operative pain (other than biliary colic) nor chronic pain conditions, nor uncontrolled chronic conditions, nor cancer, nor a laboratory abnormality that the investigator considered to contraindicate study participation
* Patient had any cognitive impairment that would, in the investigator's opinion, preclude study participation or compliance with protocol mandated procedures
* Patient had a history of known alcohol, analgesic, or narcotic substance abuse within the one year prior to Screening
* Patient had any laboratory abnormality at screening, that, in the opinion of the investigator, is not due to the condition requiring surgery and is not expected to resolve post-surgery, and would, therefore, contraindicate study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2002-11; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Patient's Global Evaluation of Study Medication | Day 2 and Day 3
Summed Pain Intensity (categorical) through 24 hours (SPI 24) | Day 2 and Day 3

SECONDARY OUTCOMES:
Time-specific PI (VAS) | Days 2 to 5
Patient's Global Evaluation of Study Medication | Day 4 and Day 5
Time to first dose of rescue medication | Days 2 to 5
Percent of patients who took rescue medication on each study day | Days 2 to 5
Amount of rescue medication taken | Days 2 to 5
Time between doses of study medication | Days 2 to 5
Worst PI (derived from the mBPI-SF) | Days 2 to 5
Average PI (derived from the mBPI-SF) | Days 2 to 5
SPI 24 (categorical) | Day 4 and Day 5
Time-specific PI (categorical) | Days 2 to 5
SPI 24 (VAS) | Days 2 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (50):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Daphne, Alabama
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Sheffield, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Woodland, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Blue Ridge, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Germantown, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Silver Spring, Maryland
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Universal City, Texas
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Suffolk, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALA-0513-145&StudyName=A%20Multiple-dose%2C%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%20Study%20of%20the%20Analgesic%20Efficacy%20and%20Safety%20of%20Valdecoxib%20Compared%20to%20